CLINICAL TRIAL: NCT04053816
Title: The TIGHT-K STUDY. Prevention of Dysrhythmias on the Cardiac Intensive Care Unit - Does Maintenance of High-normal Serum Potassium Levels Matter
Brief Title: Prevention of Dysrhythmias on the Cardiac Intensive Care Unit - Does Maintenance of High-normal Serum Potassium Levels Matter
Acronym: TIGHT-K
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Aberdeen Royal Infirmary (Other); Mid and South Essex NHS Foundation Trust (Other); Blackpool Victoria Hospital (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Derriford Hospital (Other); Deutsches Herzzentrum der Charité (Unknown); Freeman Health System (Other); Golden Jubilee National Hospital (Other Government); Guy's and St Thomas' NHS Foundation Trust (Other); Hammersmith Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); King's College Hospital NHS Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); Royal Infirmary of Edinburgh (Other); Royal Sussex County Hospital (Other); St George's University Hospitals NHS Foundation Trust (Other); Universität Münster (Other); Wythenshawe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260639
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Arrhythmias, Cardiac
Keywords: cardiovascular; potassium supplementation; cardiac surgery; atrial fibrillation; coronary artery bypass grafting; potassium
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Potassium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxed control (Experimental): Those randomised to the 'Relaxed' Group will receive potassium supplementation only if their serum potassium drops below 3.6 mEq/L.
  Interventions: Drug: Potassium
- Tight control (Active Comparator): Patients randomised to the 'Tight' group will receive potassium supplementation if their serum potassium falls below 4.5 mEq/L (current practice).
  Interventions: Drug: Potassium

INTERVENTIONS:
Drug: Potassium — The trial treatment will start when patients are admitted to the intensive care unit after their surgery. The patient will undergo regular blood investigations, as per current practice. The frequency of K+ monitoring while on ICU will be according to clinician / nursing staff preference.
  Potassium supplementation will be according to local hospital protocols. This can be either via an intravenous infusion or as a tablet. Patients will otherwise be treated as per current hospital protocol.

SUMMARY:
The purpose of this study is to determine whether a strategy of maintaining serum potassium levels at ≥3.6 mEq/L is non-inferior to a strategy of usual treatment (≥4.5 mEq/L) on the occurrence of new onset atrial fibrillation after cardiac surgery (AFACS) in patients undergoing isolated coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
At least one in three patients is affected by atrial fibrillation after cardiac surgery(AFACS), with most episodes occurring in the first five postoperative days. AF occurrence is associated with increased morbidity, short and long-term mortality, intensive care unit (ICU) and hospital stay and cost of care. Persistence of these associations after adjustment for potential confounding factors suggests that they may be causal. The incidence and prevalence of AF and its associated costs are expected to increase as the surgical population ages. Extensive effort is undertaken to prevent AF after cardiac surgery from occurring, but clinical practice in this area is highly variable and the evidence base for most interventions is sparse.

Potassium plays an important role in cardiac electrophysiology. Serum potassium concentrations ([K+]) are commonly low following cardiac surgery, and appear marginally lower in those suffering atrial arrhythmias in non-surgical cohorts. Despite an absence of proof that this association is causal, efforts to maintain serum [K+] in the 'high-normal' range (≥ 4.5 mEq/L), as opposed to just intervening if potassium drops below its lower 'normal' threshold (<3.6 mEq/L), are considered 'routine practice' for AF prevention in post-surgical patients in many centres across the world.

From the (unpublished) data from our Tight-K Feasibility Study, all 160 patients would have required at least one dose of potassium to supplement their levels to this high-normal range and 45.5% of all serum [K+] measurements were below 4.5mEq/L at some point. Data from the same pilot study show a median number of potassium doses given in the 'tight' group (high-normal serum potassium target) of seven, compared to a median of one, with most patients not receiving any potassium supplementation at all, in the 'relaxed' group. This demonstrated for the first time ever, that the practice does achieve a separation in serum potassium levels between the two groups, so the protocol is indeed effective in achieving higher serum potassium levels.

The efficacy of the practice of maintaining high-normal serum potassium levels for the prevention of AF after cardiac surgery, however, remains unproven and data supporting it are extremely limited, being derived from observational studies rather than randomised trials. Indeed, no data exist to demonstrate that maintaining a high-normal potassium level is beneficial in these circumstances, or that aggressive replenishment of potassium in these patients improves outcome.

Meanwhile, potassium supplementation may cause discomfort or harm. Routine central venous potassium administration in the early post-operative period, when oral supplementation is not possible, is time-consuming, costly and associated with clinical risk: rapid infusion can prove fatal, and leaving central venous catheters in situ for the sole purpose of potassium replacement increases infection risk. Oral replacement (when feasible) is commonly associated with profound nausea and gastrointestinal side effects, and is very poorly tolerated by patients. The annual costs of intravenous potassium exceed those for other drugs in many cardiac surgical units due to the large quantities administered. Nursing time (e.g. for drug checks and administration) will add to this cost.

The routine maintenance of serum [K+] ≥ 4.5 mEq/L is a costly practice of unproven efficacy that is unpleasant and may be hazardous for patients. The investigators shall address this issue, performing the first appropriately powered non-inferiority multicentre randomised trial of potassium supplementation in patients undergoing coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to have isolated CABG surgery
* Patient in sinus rhythm

Exclusion Criteria:

* Age less than 18 years
* Previous history of Atrial Fibrillation, Atrial Flutter and/or Atrial Tachyarrhythmia
* Pre-operative high-degree atrioventricular (AV) block (defined as Mobitz type 2 second degree AV block or complete heart block)
* Pre-operative serum [K+] greater than 5.5 mEq/L
* Current/previous use of medication for the purposes of cardiac rhythm management
* Dialysis-dependent end-stage renal failure
* Concurrent patient involvement in another clinical trial assessing cardiac rhythm post-operative interventions
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1684 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
The presence of new onset AFACS until until hour 120 after initial admission to ICU/post-operative care facility, or discharge from hospital, whichever occurs first. | Maximum of 5 days
  Episode of AFACS lasting ≥30 seconds that is both clinically detected and electrocardiographically confirmed (on either a 12-lead electrocardiogram (ECG), telemetry or Holter monitoring

SECONDARY OUTCOMES:
The incidence of new onset AFACS | Maximum of 5 days
  Detected on Holter monitor until hour 120 after initial admission to ICU/post-operative care facility or discharge from hospital, whichever occurs first.
The incidence of at least one episode of AFACS | Maximum of 5 days
  Clinically identified AFACS or Holter-identified AFACS until hour 120 after initial admission to ICU/post-operative care facility or discharge from hospital, whichever occurs first.
Number of patients experiencing at least one episode of a non-AF arrhythmia. | Maximum of 5 days
  Identified on Holter monitor until hour 120 after after initial admission to ICU/post-operative care facility or discharge from hospital, whichever occurs first
In-patient mortality | Maximum 6 months
6-month mortality | Maximum 6 months
Critical care length of stay | Maximum 6 months
  Number of days patients are in inpatients in critical care
Hospital length of stay | Maximum 6 months
  Number of days patients are inpatients in all hospital wards
Costs relating to potassium therapy | Maximum of 5 days
  Financial cost of administering potassium therapy to patients
Quality of life at 6 months: questionnaire | 6 months
  Quality of life questionnaire(EQ-5D-5L) administered before surgery and at 6 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, Sutton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] O'Brien B, Campbell NG, Allen E, Jamal Z, Sturgess J, Sanders J, Opondo C, Roberts N, Aron J, Maccaroni MR, Gould R, Kirmani BH, Gibbison B, Kunst G, Zarbock A, Kleine-Bruggeney M, Stoppe C, Pearce K, Hughes M, Van Dyck L, Evans R, Montgomery HE, Elbourne D; TIGHT K investigators. Potassium Supplementation and Prevention of Atrial Fibrillation After Cardiac Surgery: The TIGHT K Randomized Clinical Trial. JAMA. 2024 Sep 24;332(12):979-988. doi: 10.1001/jama.2024.17888. PMID 39215972
- [Derived] Campbell NG, Allen E, Evans R, Jamal Z, Opondo C, Sanders J, Sturgess J, Montgomery HE, Elbourne D, O'Brien B. Impact of maintaining serum potassium concentration >/= 3.6mEq/L versus >/= 4.5mEq/L for 120 hours after isolated coronary artery bypass graft surgery on incidence of new onset atrial fibrillation: Protocol for a randomized non-inferiority trial. PLoS One. 2024 Mar 13;19(3):e0296525. doi: 10.1371/journal.pone.0296525. eCollection 2024. PMID 38478488